CLINICAL TRIAL: NCT01788384
Title: A Multicenter, Double-blind, Randomized, Vehicle-controlled, Parallel-group Study Comparing Clindamycin Phosphate and Benzoyl Peroxide Gel and Acanya® 1.2%/2.5% and Both Active Treatments to Vehicle Control for Treating Acne Vulgaris
Brief Title: Evaluate Therapeutic Equivalence and Safety of Two Clindamycin Phosphate and Benzoyl Peroxide Gels in Acne Vulgaris
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Watson Laboratories, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 12-1001
Record Dates: First submitted 2013-02-07; First posted 2013-02-11 (Estimated); Last update posted 2013-02-11 (Estimated); Status verified 2013-02

CONDITIONS: Acne Vulgaris
Keywords: acne; Clindamycin Phosphate/Benzoyl Peroxide; Acanya; Mild to severe acne vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — clindamycin phosphate; Drugs, Generic; clindamycin phosphate benzoyl peroxide combination

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Acanya (Active Comparator): Acanya® (Clindamycin Phosphate and Benzoyl Peroxide) Gel, 1.2%/2.5% gel (Valeant Pharmaceuticals, North America)
  Interventions: Drug: Clindamycin Phosphate and Benzoyl Peroxide Gel, 1.2%/2.5%
- Clindamycin Phosphate / Benzoyl Peroxide (Experimental): Clindamycin Phosphate / Benzoyl Peroxide Gel, 1.2%/2.5%
  Interventions: Drug: Clindamycin Phosphate / Benzoyl Peroxide Gel
- Vehicle Gel (Placebo Comparator): Placebo (Vehicle Gel)of the test product (Watson Laboratories, Inc.)
  Interventions: Drug: Placebo (Vehicle Gel)

INTERVENTIONS:
Drug: Clindamycin Phosphate / Benzoyl Peroxide Gel — Dosage form: topical gel Dosage: One pea-sized amount will be applied onto six areas of the face (chin, left cheek, right cheek, nose, left forehead, right forehead), avoiding the eyes, lips and mucous membranes.
  Other Names: Generic
  Arms: Clindamycin Phosphate / Benzoyl Peroxide
Drug: Clindamycin Phosphate and Benzoyl Peroxide Gel, 1.2%/2.5% — Dosage form: topical gel Dosage: One pea-sized amount will be applied onto six areas of the face (chin, left cheek, right cheek, nose, left forehead, right forehead), avoiding the eyes, lips and mucous membranes.
  Other Names: Acanya
  Arms: Acanya
Drug: Placebo (Vehicle Gel) — Dosage form: topical gel Dosage: One pea-sized amount will be applied onto six areas of the face (chin, left cheek, right cheek, nose, left forehead, right forehead), avoiding the eyes, lips and mucous membranes.
  Other Names: Vehicle Gel
  Arms: Vehicle Gel

SUMMARY:
Acanya (Clindamycin Phosphate and Benzoyl Peroxide) Gel, 1.2%/2.5% gel marketed by Valeant Pharmaceuticals, North America, is a safe and effective topical therapy used for the treatment of acne vulgaris.

DETAILED DESCRIPTION:
Watson Laboratories, Inc. has developed a generic formulation of Clindamycin Phosphate and Benzoyl Peroxide Gel, 1.2%/2.5%,and the current study is designed to evaluate the safety and efficacy of this formulation to determine if it is bioequivalent to Acanya.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or non pregnant female
* ≥ 12 and ≤ 40 years
* Diagnosis of acne vulgaris (acne)
* >18 years and provide written informed consent
* Ages 12 to 17 and provide written assent and written informed consent from patient's legal representative
* Must sign a HIPAA authorization
* Minimum ≥ 25 non-inflammatory lesions
* ≥ 20 inflammatory lesions
* ≤ 2 nodulocystic lesions on the face
* Acne of severity grade 2, 3, or 4 -Investigator's Global Assessment (IGA)
* Refrain from all other topical acne medications or antibiotics during the 12-week treatment period except Investigational Product
* All Female patients with a negative urine pregnancy test who use birth control from the study start to 30 days after the last administration of study drug
* All male patients who use birth control with their partners, from the study start to 30 days after the last administration of study drug. Abstinence is acceptable. Female partners should use birth control
* Must be willing and able to understand and comply with the protocol requirements and required study visits
* In good health
* Free from any clinically significant disease
* Must have used the same brands/types of make-up for a minimum period of 14 days prior to study entry and must agree to use the same make-up, brand/type and maintain the same frequency of use throughout the study

Exclusion Criteria:

* Female patients who are pregnant, nursing or planning to become pregnant during study
* History or presence of Crohn's disease, ulcerative colitis, regional enteritis, or antibiotic-associated colitis
* Hypersensitivity or allergy to benzoyl peroxide, clindamycin and/or any of the study medication ingredients
* Presence of any skin condition that would interfere with the diagnosis or assessment
* Excessive facial hair
* Wax epilation of the face within 14 days prior
* Used oral retinoids or therapeutic vitamin A supplements of >10,000 units/day (multivitamins are allowed) within 6 months prior to or during the study
* Estrogens or oral contraceptives for <3 months prior to baseline; Use of such therapy must remain constant throughout the study
* Cryodestruction, chemodestruction, dermabrasion, photodynamic therapy, acne surgery, intralesional steroids, X-ray therapy procedures performed on the face within 1 month prior to or during the study
* Any systemic (steroids, antibiotics treatment for acne, anti-inflammatory agents) treatments within 1 month prior to baseline or during the study
* Any (topical steroids, topical retinoids, α-hydroxy/glycolic acid, benzoyl peroxide, topical anti-inflammatory agents, topical antibiotics) treatments within 2 weeks prior to baseline or during the study:
* Intend to use Spironolactone
* Intend to use tanning booths, sunbathing, or excessive exposure to the sun
* Radiation therapy and/or anti-neoplastic agents within 90 days prior to baseline
* Unstable clinically significant medical disorders or life-threatening diseases
* On-going malignancies requiring systemic treatment
* Any malignancy of the facial area skin
* Engage in activities that involve excessive or prolonged exposure to sunlight or weather extremes
* Consume excessive amounts of alcohol or use drugs of abuse
* Participation in an investigational drug study within 30 days prior
* Are participating in non-treatment studies such as observational studies or registry studies can be considered for inclusion
* Previously enrolled in this study
* Laser therapy, electrodessication and phototherapy to the facial area within 180 days prior to study entry
* Cosmetic procedures which may affect the efficacy and safety profile of the study drug within 14 days prior to study entry
* Currently have or have recently had bacterial folliculitis on the face

Ages: 12 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 708 (Actual)
Dates: Start 2012-07; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
The evaluation of the primary endpoint will be based on the mean percent changes from baseline to week 12 in the inflammatory (papules and pustules) lesion counts and in the non-inflammatory (comedones) lesion counts. | Week 12

SECONDARY OUTCOMES:
The proportion of subjects with a clinical response of "success" at Week 12 using IGA. | 12 Weeks
  The proportion of subjects with a clinical response of "success" at Week 12. Success was defined as an IGA score that was at least 2 grades less than the baseline assessment.

OTHER OUTCOMES:
Analysis of Application Site Reactions | 12 Weeks
  A descriptive analysis comparing the application site reactions for each treatment group will be conducted to ensure that the test product is not worse than the reference product with regard to the expected and unexpected application site reactions.
Safety analyses were conducted on the Safety population. | 12 Weeks
  Safety incidence of all AEs reported during the study was summarized using the Medical Dictionary for Drug Regulatory Activities (MedDRA), by treatment group, body system, severity, and relationship to study drug.
  The report of AEs included date of onset, description of the AE, and date of resolution.

CONTACTS AND LOCATIONS:
Overall Officials: John L Capicchioni, Study Director — Akesis, LLC